CLINICAL TRIAL: NCT05490290
Title: Medical Imaging Decision And Support
Acronym: MIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Collaborators: Erasmus Medical Center (Other); University Hospital Schleswig-Holstein (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SFV-89-19
Record Dates: First submitted 2022-06-29; First posted 2022-08-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Clinical Decision Support Systems
Keywords: Diagnostic Imaging; Referral; Healthcare Costs; Guidelines as Topic; Clinical Trial Protocol; Overdiagnosis; Radiology
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will be performed as a multi-center cluster randomized trial with departments acting as clusters combined with a before-after-revert design. Four hospitals with each 8 participating departments for a total of 32 clusters will be included in the study. All departments will start with the control condition. Subsequently, stratified per specialty (surgical vs. non-surgical), half of the departments - chosen at random - will switch to the active intervention while the other remain in the control condition.
  Amendments November 2023:
  I)see Study Description
  II) We made an amendment to the applied sample size calculation. The original sample size for MERC review was calculated using clusterPower version 0.6.111 function crtpwr.2prop. The amended sample size calculation that in the online publication of the protocol applies a newer, more appropriate version of clusterPower version 0.7.0 using the function cpa.did.binary.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): In the active intervention the CDSS is implemented with decision support. Physicians are made aware of the referral guidelines and appropriate exams are suggested. Their imaging requests are categorized as appropriate, under certain conditions appropriate, or inappropriate and feedback is provided. Physicians are able to change their request in response to the feedback.
  Interventions: Other: Active
- Control (No Intervention): The control condition will consist of computerized order entry with structured data entry of the clinical indication and tracking of the imaging exams requested. The CDSS is implemented but without decision support and physicians are blinded to these referral guidelines. Without their knowledge their imaging requests are categorized as appropriate, under certain conditions appropriate, or inappropriate. They receive no feedback to their requests.

INTERVENTIONS:
Other: Active — In the active intervention condition, decision support is provided during the referral procedure of medical imaging exams.
  Arms: Active

SUMMARY:
Rationale: Diagnostic medical imaging is essential in health care and guides patient management decisions. Rapid advances in imaging technology have enabled diagnosis at an early disease stage. Nevertheless, striving for early diagnosis leads to substantial overuse of diagnostic tests (too many tests are performed) and overdiagnosis (diagnosed abnormalities that are unlikely to affect a patient's health or well-being), with dire consequences to patient outcomes and health care costs. Computerized decision support systems (CDSS), such as the European Society of Radiology (ESR) iGuide, have been developed to guide referring physicians at the point of care. Objective: The overall objective of this project is to promote the appropriate, meaningful, value-based and personalized use of medical imaging. The specific objectives of this study are to evaluate the trends over time with implementation of a CDSS to guide imaging referrals (ESR iGuide) in key outcomes related to the appropriate use of diagnostic imaging tests, and to compare these trends between departments randomized between implementation of the active intervention (with decision support) and the control condition (no decision support). Study design: The study will be performed as a multi-center cluster randomized trial with departments acting as clusters combined with a before-after-revert design. Four hospitals with each 8 participating departments for a total of 32 clusters will be included in the study. All departments will start with the control condition. Subsequently, stratified per specialty (surgical vs non-surgical), half of the departments - chosen at random - will switch to the active intervention while the other half in the control condition. Study population: The study population consists of patients of eligible participating departments for whom a diagnostic imaging procedure is considered, and for whom a diagnostic imaging request is entered in a computerized order entry in such a form that it is registered by the CDSS.

Intervention: The control condition will consist of computerized order entry with structured data entry of the clinical indication and tracking of the imaging exams requested. The CDSS is implemented but without decision support and physicians are blinded to these referral guidelines. Without their knowledge their imaging requests are categorized as appropriate, under certain conditions appropriate, or inappropriate. They receive no feedback to their requests. In the active intervention the CDSS is implemented with decision support. Physicians are made aware of the referral guidelines and appropriate exams are suggested. Their imaging requests are categorized as appropriate, under certain conditions appropriate, or inappropriate and feedback is provided. Physicians are able to change their request in response to the feedback. In the revert condition decision support is removed to study the sustainable educational effect of temporary use of the system. Main study parameters/endpoints: The primary outcome is the proportion of inappropriate diagnostic imaging exams requested per cluster (department). Inappropriateness is determined by the decision support system and is based on the ESR imaging referral guidelines. Secondary outcomes are the overall absolute number of imaging exams ordered (total and by exam type), estimated medical radiation from diagnostic imaging in investigated groups, and estimated medical costs for diagnostic imaging from the healthcare system perspective in investigated groups.

Amendment November 2023:

At Johannes Gutenberg University Mainz, the CDSS could not be integrated into the hospital's internal computerized order entry system as required for the study. Therefore, departments from this hospital were not eligible for inclusion. Therefore, and 24 instead of 32 departments were from three locations (Augsburg, Kiel, Lübeck) were randomized accordingly. In a qualitative description of the process of integrating the CDSS in the local hospitals, Mainz will still be included.

ELIGIBILITY:
Inclusion Criteria:

• Departments in hospitals that were able to integrate the ESR iGuide system in the ordering system

Exclusion Criteria:

• Departments without electronic medical records or without integration of the decision support system into their computerized order entry system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Appropriateness of diagnostic imaging exams | 1 year
  The primary outcome is the proportion of inappropriate diagnostic imaging exams in total exams requested per cluster (department) measured by ESR iGuide report tool.

SECONDARY OUTCOMES:
Absolute number of imaging exams | 1 year
  Overall absolute number of imaging exams ordered, total and by exam type.
Medical radiation from diagnostic imaging | 1 year
  For all types of exams performed the average radiation dose will be collected and multiplied by the number of those types of exams performed.
Medical costs for diagnostic imaging | 1 year
  For all types of exams performed the average costs (German costs, healthcare perspective) will be determined and multiplied by the number of those types of exams performed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kroencke T, Dijk SW, Halfmann MC, Wollny C, Barkhausen J, Janssen O, Rizopoulos D, Myriam Hunink MG. Challenges and insights from implementing clinical decision support systems for radiologic imaging: experience from the MIDAS trial. Insights Imaging. 2025 Jul 5;16(1):152. doi: 10.1186/s13244-025-02027-0. PMID 40616704
- [Derived] Dijk SW, Wollny C, Barkhausen J, Jansen O, Mildenberger P, Halfmann MC, Stroeder J, Rizopoulos D, Hunink MGM, Kroencke T. Evaluation of a Clinical Decision Support System for Imaging Requests: A Cluster Randomized Clinical Trial. JAMA. 2025 Apr 8;333(14):1212-1221. doi: 10.1001/jama.2024.27853. PMID 39928308
- [Derived] Dijk SW, Kroencke T, Wollny C, Barkhausen J, Jansen O, Halfmann MC, Rizopoulos D, Hunink MGM. Medical Imaging Decision And Support (MIDAS): Study protocol for a multi-centre cluster randomized trial evaluating the ESR iGuide. Contemp Clin Trials. 2023 Dec;135:107384. doi: 10.1016/j.cct.2023.107384. Epub 2023 Nov 8. PMID 37949165
- See also: Study Protocol Published in the journal Contemporary Clinical Trials - "Medical Imaging Decision And Support (MIDAS): Study protocol for a multi-centre cluster randomized trial evaluating the ESR iGuide" — http://doi.org/10.1016/j.cct.2023.107384